CLINICAL TRIAL: NCT00521703
Title: Evaluation of Topical Lidocaine Spray as Adjuvant to Upper Gastrointestinal Endoscopy in Children and Teenagers
Brief Title: Evaluation of Topical Lidocaine Spray as Adjuvant to Upper Gastrointestinal Endoscopy in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Infantil Cândido Fontoura (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HICF 001-07
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Dyspepsia; Malabsorption Syndrome; Gastroesophageal Reflux Disease; Abdominal Pain
Keywords: endoscopy, gastrointestinal; lidocaine; propofol; child; adolescent
MeSH Terms: conditions — Dyspepsia; Malabsorption Syndromes; Gastroesophageal Reflux; Abdominal Pain | interventions — Lidocaine; tannic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): group treated
  Interventions: Drug: Lidocaine
- 2 (Placebo Comparator): control group
  Interventions: Drug: Tannic acid

INTERVENTIONS:
Drug: Lidocaine — oral cavity and throat were sprayed with lidocaine 10% two to three puffs before propofol infusing
  Arms: 1
Drug: Tannic acid — oral cavity and throat were sprayed with placebo (tannic acid 0.5%) two to three puffs before propofol infusing
  Arms: 2

SUMMARY:
There is some controversy in the medical literature regarding the effectiveness of topical lidocaine in children as an adjuvant drug to upper gastrointestinal endoscopy. In children, deep sedation and general anesthesia are often used to sedate children submitting to this procedure. Propofol is an anesthetic drug increasingly popular in this situation, but this drug can only be used with an anesthesiologist in Brazil. Its main side effects include hypotension, respiratory depression and local pain. Lidocaine is frequently used as premedication, and the rationale is that lowering patient discomfort could lower the required dose to achieve the endoscopy and reduce potential side effects. Nevertheless, some patients perceive this medication as uncomfortable. This study aims to compare sedative drug doses between patients who were given either placebo or topical lidocaine.

DETAILED DESCRIPTION:
This study is a randomized double-blind placebo-controlled clinical trial.

Primary outcome: propofol doses required to achieve adequate sedation.

Population: children submitting to upper digestive endoscopy, weight > 30 kg and age between 8 and 18 years.

Exclusion criteria: neurological disorders, psychiatric disorders, specific contra-indication to either lidocaine or propofol.

Estimated sample: 160 patients. Placebo: tannic acid 0.5%

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents submitting to upper digestive endoscopy with weight above 30 kg and age between 8 and 18 years

Exclusion Criteria:

* Neurological disorders
* Psychiatric disorders
* Specific contra-indication to lidocaine
* Specific contra-indication to propofol

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2007-08; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
propofol dose required to achieve adequate sedation to upper digestive endoscopy | one hour

SECONDARY OUTCOMES:
incidence of tachycardia (heart rate > 120) during the procedure | one hour
incidence of hypoxemia (SpO2 < 94%) during procedure | one hour
severity of sore throat after the procedure | up to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Machado, PhD, Principal Investigator — UNIFESP/EPM
Locations (1):
- Hospital Infantil Cândido Fontoura, São Paulo, São Paulo, Brazil